CLINICAL TRIAL: NCT03554434
Title: An Expanded Access Program for AM0010 (Pegilodecakin) Subcutaneous Injection
Brief Title: An Expanded Access Program for AM0010 (Pegilodecakin)
Status: No longer available | Type: Expanded Access
Sponsor: Eli Lilly and Company (Industry)
Collaborators: ARMO BioSciences (Industry)
Responsible Party: Sponsor
Other Study IDs: AM0010-99
Record Dates: First submitted 2018-05-31; First posted 2018-06-13 (Actual); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Melanoma; Prostate Cancer; Ovarian Cancer; Renal Cell Carcinoma; Colorectal Carcinoma; Pancreatic Carcinoma; Non-small Cell Lung Carcinoma; Solid Tumors; Breast Cancer
MeSH Terms: conditions — Melanoma; Prostatic Neoplasms; Ovarian Neoplasms; Carcinoma, Renal Cell; Colorectal Neoplasms; Pancreatic Neoplasms; Carcinoma, Non-Small-Cell Lung; Breast Neoplasms | interventions — AM0010; pegilodecakin

INTERVENTIONS:
Biological: AM0010 — AM0010
  Other Names: LY3500518; Pegilodecakin

SUMMARY:
This is an Expanded Access Program (EAP) available to patients who have advanced cancers, who have failed or progressed on standard of care systemic therapy and do not qualify for ongoing clinical trials.

ELIGIBILITY:
* Patient is NOT eligible for other AM0010 clinical trials currently open in the region
* Patient is in urgent need of therapy who fail to meet eligibility criteria for other clinical trials related to AM0010 (PEG-IL-10) can be considered for enrollment into this Expanded Access Program.
* Patient has advanced cancer in indications where preliminary anti-tumor efficacy of AM0010 has been demonstrated or where AM0010 mediated immune activation is likely to benefit the patient.
* Patient has failed or progressed on standard of care (SOC) systemic therapy
* Patient is refusing SOC therapy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Contact Lilly at 1-800-LillyRx (1-800-545-5979), Study Director — Eli Lilly and Company